CLINICAL TRIAL: NCT03463278
Title: The Impact of Blastulation Rate in the Outcome of Freeze All Strategy: COMFFETI Trial, Cumulative Delivery Rate
Brief Title: The Number of Blastocysts Formed in the Outcome of Freeze All Strategy: COMFFETI Trial, Cumulative Delivery Rate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assisting Nature (Other)
Responsible Party: Sponsor
Other Study IDs: Blastocyst-AN004
Record Dates: First submitted 2018-03-02; First posted 2018-03-13 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy, Ovarian
Keywords: blastocyst; Freeze-all; IVF; Cumulative results; cumulative delivery rate
MeSH Terms: conditions — Pregnancy, Ovarian | interventions — Pregnancy Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 0-4 blastocysts: group A: cumulative pregnancy rate of 0-4 blastocysts vitrified
  Interventions: Diagnostic Test: Pregnancy Rate
- 5-7 blastocysts: group B: cumulative pregnancy rate of 5-7 blastocysts vitrified
  Interventions: Diagnostic Test: Pregnancy Rate
- >7 blastocysts: group C: cumulative pregnancy rate of >7 blastocysts vitrified
  Interventions: Diagnostic Test: Pregnancy Rate

INTERVENTIONS:
Diagnostic Test: Pregnancy Rate — The pregnancy and live birth rate according to number of blastocysts formed in our three groups

SUMMARY:
A prospective study of the blastulation rate in the outcome of the Freeze all strategy

DETAILED DESCRIPTION:
A prospective study of the blastulation rate in women under the age of 40 years following Freeze all strategy, according to AMH levels and sperm parameters.

Study group 1: number of vitrified blastocysts 0-4 Study group 2: number of vitrified blastocysts 5-7 Study group 3: number of vitrified blastocysts >7

ELIGIBILITY:
Inclusion Criteria:

* primary infertility
* age 20-39 years;
* body mass index (BMI) 18-29kg/m2;
* regular menstrual cycle of 26-35days,
* presumed to be ovulatory;
* >1mil/ml spermatozoa;
* short antagonist protocol

Exclusion Criteria:

* poor responders;
* age ≥40;
* TESE sperm;
* PGS cycles;
* donor oocytes;
* donor sperm

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged 20-39 years old following blastocyst culture after ICSI cycle in Freeze all Strategy
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2013-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative Live Birth rate according to blastulation rate | 5 days of embryo culture
  Cumulative Live Birth rate according to blastulation rate

SECONDARY OUTCOMES:
Cumulative Pregnancy rate according to blastulation rate | 5 days of embryo culture
  Cumulative Pregnancy rate according to blastulation rate

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Papanikolaou, MD, PhD, Principal Investigator — Assisting Nature
Locations (1):
- Assisting Nature, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided